CLINICAL TRIAL: NCT05435118
Title: Use of the Equimolar Mixture of Oxide Nitrous and Oxygen (EMONO) Associated With Audiovisuals During Peripheral Venous Access Insertion of Children Between 2-5 Years Old Children
Brief Title: Use of the Equimolar Mixture of Oxide Nitrous and Oxygen (EMONO) Associated With Audiovisuals in Children
Acronym: EMONO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale di Lodi (Other)
Responsible Party: Principal Investigator, Stefano Maiandi, MSc PhDs - Health Professionals Directorate, Azienda Socio Sanitaria Territoriale di Lodi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INF202201
Record Dates: First submitted 2022-05-27; First posted 2022-06-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pain, Acute; Child, Only; Nurse's Role; Nitrous Oxide
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMONO (usual care administered to all the children undergoing painful procedures) (No Intervention): Use of the Equimolar Mixture of Oxide Nitrous and Oxygen (EMONO) with facial mask. In the hospital EMONO is administered to all the children for procedure pain control.
- EMONO + audiovisuals tool (Experimental): Use of the Equimolar Mixture of Oxide Nitrous and Oxygen (EMONO) with facial mask and vision of audiovisual toll with smartphone or tablet. The intervention is represented by the audiovisual tool.
  Interventions: Other: EMONO + audiovisuals tool

INTERVENTIONS:
Other: EMONO + audiovisuals tool — EMONO + use of audiovisuals tool on smartphone or tablet
  Arms: EMONO + audiovisuals tool

SUMMARY:
Children experience numerous painful experiences from nursing procedures: peripheral venous access placement is the main cause of procedural pain.

As much as pharmacological and nonpharmacological tools are known, their application during venipuncture is not systematic by children's hospitals.

Among pharmacological tools, the Equimolar Mixture of Nitrogen Protoxide and Oxygen (EMONO) provides adequate protection from procedural pain through inhalation of the gas mixture at least 3 minutes before the procedure.

Literature reports that the combination of nonpharmacological distractive tools and pharmacological interventions increases their analgesic effect.

The aim of the study is to measure children's cooperation during procedure (primary outcome), pain perception and side effects when EMONO is combined with audiovisuals compared with EMONO alone in peripheral venous access placement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 years and 5 years and 364 days
* Prescription for peripheral venous access placement
* Parental consent for participation in the study
* Presence of at least one parent in possession of a smartphone/tablet with the ability to connect to the Internet through Wi-Fi available to users
* Absence of contraindications to the administration of EMONO reported in health records
* Absence of facial pathology
* Presence on duty of at least one experimental nurse trained in the use of EMONO

Exclusion Criteria:

* Age less than 2 years and more than 5 years and 364 days
* No parental consent to participate in the study
* Parents not in possession of a smartphone/tablet with the ability to connect to the internet through Wi-Fi available to users
* Presence of contraindications to EMONO administration
* Presence of facial pathology
* Oxygen therapy
* Presence of tracheostomy
* Absence on duty of at least one experimental nurse trained in the use of EMONO

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
collaboration | 30 minutes
  children cooperation during procedure assessed with Groningen Distress Rating Scale (Humphrey et al., 1992; Herd et al., 2006; Doumit et al., 2016)

SECONDARY OUTCOMES:
pain perception in 2 years-old children | 30 minutes
  pain perceprion during procedure assessed with FLACC scale (Merkel et al., 1997)
pain perception in 3 to 5 years-old children | 30 minutes
  pain perceprion during procedure assessed with Wong-Baker scale (Wong and Baker, 1988)
side effect 1 | 30 minutes
  vomiting during procedure Due to not available scales, numerical values from 0 (absence of sign) to 3 (presence of sign requiring medical intervention ) will be assigned to these signs
side effect 2 | 30 minutes
  gag reflex during procedure Due to not available scales, numerical values from 0 (absence of sign) to 3 (presence of sign requiring medical intervention ) will be assigned to these signs

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Maiandi, PhDs, Principal Investigator — Azienda Socio Sanitaria Territoriale di Lodi
Locations (1):
- Stefano Maiandi, Lodi, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maiandi S, Coluccia S, Ghizzardi G, Nicardi R, Giacchero R, Lusignani M, Gianni ML, Edefonti VC. Effectiveness of Equimolar Mixture of Oxygen and Nitrous Oxide Combined With Audiovisual in Young Children: A Randomised Controlled Trial. Eur J Pain. 2025 Sep;29(8):e70096. doi: 10.1002/ejp.70096. PMID 40762409
- [Derived] Maiandi S, Ghizzardi G, Edefonti V, Giacchero R, Lusignani M, Gianni ML. Is the equimolar mixture of oxygen and nitrous oxide (EMONO) associated with audiovisuals effective in reducing pain and side effects during peripheral venous access placement in children? Protocol for a single-centre randomised controlled trial from Italy. BMJ Open. 2023 Jul 7;13(7):e067912. doi: 10.1136/bmjopen-2022-067912. PMID 37419632